CLINICAL TRIAL: NCT00187213
Title: Biventricular Versus Left Univentricular Pacing With ICD Back-up in Heart Failure Patients
Brief Title: B-Left HF: Biventricular Versus Left Univentricular Pacing With Implantable Cardiac Defibrillator (ICD) Back-Up in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Christophe Bailleul, St. Jude Medical
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR03019HF
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; Ventricular Dysfunction; Heart Diseases
Keywords: Ventricular Dyssynchrony
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Heart Diseases | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy

SUMMARY:
The purpose of this study is to demonstrate that biventricular pacing (BiV) and left univentricular (left ventricular [LV] only) pacing are safe and effective for cardiac resynchronization therapy in heart failure patients implanted with a cardiac resynchronization therapy defibrillator (CRT-D) device.

The hypothesis to be tested by this clinical investigation is that patients indicated for an ICD with cardiac resynchronization therapy respond as well to LV only pacing as to BiV pacing.

ELIGIBILITY:
Inclusion Criteria:

* Have an approved indication for implantation of an ICD for treatment of a life-threatening ventricular tachyarrhythmia(s)
* Have advanced heart failure with a New York Heart Association (NYHA) classification of III or IV, despite receiving a minimum of 30 days of stable optimal pharmacological therapy
* Have a ventricular conduction delay manifested as a QRS width >= 130 ms
* Have a left ventricular end diastolic diameter (LVEDD) >= 55 mm
* Have a left ventricular ejection fraction (LVEF) <= 35%

Exclusion Criteria:

* Have a CRT device already implanted
* Have a standard indication for bradycardia pacing
* Have a history of chronic atrial fibrillation [AF] (continuous AF lasting > 1 month) within 1 year prior to enrollment or have undergone cardioversion for AF in the past month)
* Have the ability to walk > 450 meters during the 6-minute walk test
* Have uncorrected primary valvular disease
* Have had a recent myocardial infarction, unstable angina or cardiac revascularization (percutaneous transluminal coronary angioplasty [PTCA] or coronary artery bypass graft [CABG]) within 1 month of enrollment
* Have had cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 3 months of enrollment
* Have a life expectancy of less than one year
* Are unable to comply with the follow-up schedule and tests
* Are minors (age below 18 years)
* Are pregnant or are planning for pregnancy in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to demonstrate that left univentricular pacing is equivalent to biventricular pacing in improving the functional capacity and inducing reverse remodeling.

SECONDARY OUTCOMES:
The secondary objective of this clinical investigation is to evaluate the proportion of improved patients in each group, using the Heart Failure Clinical Composite Response.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Leclercq, MD, PhD, Principal Investigator — CHU Pontchaillou Rennes France
Locations (1):
- Department of Cardiology - CHU Pontchaillou, Rennes, France

REFERENCES:
- [Derived] Boriani G, Kranig W, Donal E, Calo L, Casella M, Delarche N, Lozano IF, Ansalone G, Biffi M, Boulogne E, Leclercq C; B-LEFT HF study group. A randomized double-blind comparison of biventricular versus left ventricular stimulation for cardiac resynchronization therapy: the Biventricular versus Left Univentricular Pacing with ICD Back-up in Heart Failure Patients (B-LEFT HF) trial. Am Heart J. 2010 Jun;159(6):1052-1058.e1. doi: 10.1016/j.ahj.2010.03.008. PMID 20569719